CLINICAL TRIAL: NCT00321152
Title: A Double-Blind, Placebo Controlled Study of 6(S)-5-MTHF Among SSRI-Resistant Outpatients With Major Depressive Disorder (MDD)
Brief Title: A Study of 6(S)-5-MTHF Among Serotonin Reuptake Inhibitor(SSRI)-Resistant Outpatients With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pamlab, L.L.C. (Industry)
Responsible Party: George Papakostas, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006P000604
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Deplin/Deplin = participants will receive 7.5 mg/day of Deplin (6(S)-5-MTHF)for the first 4 weeks, and then 15 mg/day of Deplin for the next 4 weeks.
  Interventions: Other: 6(S)-5-MTHF (a Medical Food)
- 2 (Experimental): placebo/Deplin = participants will receive placebo for the first 4 weeks, and then 7.5 mg/day of Deplin (6(S)-5-MTHF) for the next 4 weeks.
  Interventions: Other: 6(S)-5-MTHF (a Medical Food)
- 3 (Placebo Comparator): placebo/placebo = both tablets of study medication will be placebo during both phases of the study.
  Interventions: Other: 6(S)-5-MTHF (a Medical Food)

INTERVENTIONS:
Other: 6(S)-5-MTHF (a Medical Food) — The study consists of 8 visits over a period of 8 weeks or 60 days. Eligible participants will be randomized to double-blind treatment with placebo or Deplin (6(S)-5-MTHF). Participants will have a greater than 50% chance of receiving active medication (Deplin) at some point in the 8 week study. At the end of the double-blind phase, both responders and non-responders who have completed the 8 week study will have the option of receiving free, open-label adjunctive treatment with either 7.5 mg or 15 mg of 6(S)-5-MTHF for 12 months. Subjects who agree to receive open-label treatment with 6(S)-5-MTHF for 12 months will be assessed every three (3) months until the end of the follow-up phase.

SUMMARY:
The purpose of the study is to test whether oral 6(S)-5-MTHF (Deplin®) is safe and effective in relieving depression when it is added to standard kinds of antidepressants called serotonin reuptake inhibitors (SSRIs).

DETAILED DESCRIPTION:
The study consists of two sequential phases, each lasting a total of four weeks (8 weeks total), with visits every 10 days. Once patients agree to participate in the study by signing the informed consent document, a full medical and psychiatric history will be taken and a physical examination and blood draw will be performed. Screen rating scales will be performed. Screened and eligible patients will be asked to return two weeks later for a baseline visit when they will be randomized to double-blind treatment with placebo or Deplin (6(S)-5-MTHF). The double-blind treatment will last 60 days, during which patients will be seen every 10 days. Subjects will be randomized to one of three treatment groups: a)Deplin/Deplin, b) placebo/Deplin, c) placebo/placebo. Patients will have a greater than 50% chance of receiving active medication (Deplin) at some point in the 8 week study

* For patients randomly assigned to the Deplin/Deplin sequence, the dose of 6(S)-5-MTHF will be 7.5 mg/day during the first phase of the study, and 15 mg/d during the second phase of the study.
* For patients randomly assigned to the placebo/Deplin sequence, the dose of 6(S)-5-MTHF will be 7.5 mg/day during the second phase of the study.
* For patients randomly assigned to the placebo/placebo sequence, both tablets of study medication will be placebo during both phases of the study.

All patients will be asked to take two tablets of blinded study medication in the morning, in addition to their stable dose of ongoing SSRI treatment. Each study medication tablet will be either 7.5 mg of 6(S)-5-MTHF or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Meet criteria for current Major Depressive Disorder
* Currently taking an SSRI

Exclusion Criteria:

* Pregnant women
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
* Prior course of MTHF augmentation, or intolerance to MTHF at any dose
* substance use disorders active within the last six months, any bipolar disorder (current or past), or any psychotic disorder (current or past).
* Have failed more than 2 adequate antidepressant trials during the current Major Depressive Episode.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
HAM-D | every visit

SECONDARY OUTCOMES:
QIDS-SR | every visit

CONTACTS AND LOCATIONS:
Overall Officials: George I Papakostas, M.D, Principal Investigator — Massachusetts General Hospital
Locations (11):
- United States (11):
  - University of California San Diego School of Medicine, San Diego, California
  - Rush University Medical Center, Psychiatric Medicine Associates, LLC, Chicago, Illinois
  - Lousiana State University Health Sciences Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Burlington Medical Associates, Burlington, Massachusetts
  - Waltham Family Practice, Waltham, Massachusetts
  - Charles River Medical Associates, Westborough, Massachusetts
  - Univeristy of Cincinnati, College of Medicine, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Southeast Health Consultants, LLC, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Zajecka JM, Fava M, Shelton RC, Barrentine LW, Young P, Papakostas GI. Long-term efficacy, safety, and tolerability of L-methylfolate calcium 15 mg as adjunctive therapy with selective serotonin reuptake inhibitors: a 12-month, open-label study following a placebo-controlled acute study. J Clin Psychiatry. 2016 May;77(5):654-60. doi: 10.4088/JCP.15m10181. PMID 27035404
- [Derived] Papakostas GI, Shelton RC, Zajecka JM, Etemad B, Rickels K, Clain A, Baer L, Dalton ED, Sacco GR, Schoenfeld D, Pencina M, Meisner A, Bottiglieri T, Nelson E, Mischoulon D, Alpert JE, Barbee JG, Zisook S, Fava M. L-methylfolate as adjunctive therapy for SSRI-resistant major depression: results of two randomized, double-blind, parallel-sequential trials. Am J Psychiatry. 2012 Dec;169(12):1267-74. doi: 10.1176/appi.ajp.2012.11071114. PMID 23212058